CLINICAL TRIAL: NCT02674828
Title: Physical Activity and Glycemic Control in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1509016461; DP3DK097705 (NIH)
Record Dates: First submitted 2016-01-19; First posted 2016-02-05 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reinforcement treatment (Experimental): Participants in this condition will receive reinforcement for meeting targeted physical activity goals. These subjects will receive the same treatment as standard treatment group, including incentives for uploading/synching and discussions of ADA recommendations of managing diabetes in the context of physical activity. The only difference between conditions is that participants in this condition will earn tangible reinforcement for walking the target number of steps per day (6,000 per day in week 1, 8,000 per day in week 2 and 10,000 per day in weeks 3-12). At each upload, participants will earn incentives for each day on which they met the step goals. In addition, for each 7-day period in which they meet goals on at least 5 days, they will earn bonuses.
  Interventions: Behavioral: Reinforcement for meeting targeted physical activity goals; Other: Standard of Care
- Standard Treatment (Active Comparator): Participants in the standard of care group will be told to wear Fitbit daily for 12 weeks. They will be instructed to upload or synch it >2x/week, on set days, e.g., Mon and Thurs, for the next 6 weeks and then weekly in the last 6 weeks. They will receive incentives for each upload, plus a bonus for each week in which data are registered for all 7 days in the week as scheduled. They will be encouraged to review Fitbit steps daily and on each upload/synch day. After each upload, research staff will congratulate patients via email or text for days on which they met goals, and encourage meeting goals in the upcoming week.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Reinforcement for meeting targeted physical activity goals — Participants in this condition will receive reinforcement for meeting targeted physical activity goals. These subjects will receive the same treatment as standard treatment group, including incentives for uploading/synching and discussions of ADA recommendations of managing diabetes in the context of physical activity. The only difference between conditions is that participants in this condition will earn tangible reinforcement for walking the target number of steps per day (6,000 per day in week 1, 8,000 per day in week 2 and 10,000 per day in weeks 3-12). At each upload, participants will earn incentives for each day on which they met the step goals. In addition, for each 7-day period in which they meet goals on at least 5 days, they will earn bonuses.
  Arms: Reinforcement treatment
Other: Standard of Care — Participants in the standard of care group will be told to wear Fitbit daily for 12 weeks. They will be instructed to upload or synch it >2x/week, on set days, e.g., Mon and Thurs, for the next 6 weeks and then weekly in the last 6 weeks. They will receive incentives for each upload, plus a bonus for each week in which data are registered for all 7 days in the week as scheduled. They will be encouraged to review Fitbit steps daily and on each upload/synch day. After each upload, research staff will congratulate patients via email or text for days on which they met goals, and encourage meeting goals in the upcoming week.

SUMMARY:
The purpose of this pilot study is to evaluate the initial efficacy of a reinforcement intervention to enhance physical activity levels in sedentary adolescents and young adults with type 1 diabetes (T1D). The intervention will reinforce patients for meeting physical activity goals, with escalating reinforcers provided when patients achieve continuous weeks of meeting goals. A 12-week trial will be conducted in which 60 patients will be randomized to: (1) standard care or (2) standard care plus reinforcement.

DETAILED DESCRIPTION:
Specific aims are:

1. To determine if the reinforcement intervention increases walking. The proportion of days on which participants meet walking goals will be assessed via Fitbit, a commercially available activity monitor, as well as continuous weeks on which goals are met. The hypothesis is that patients assigned to the reinforcement intervention will meet walking goals on a higher proportion of days and have longer durations of meeting walking goals than patients assigned to standard care.
2. To assess if the intervention reduces A1c. Patients randomized to the reinforcement intervention are expected to have greater decreases in A1c than patients in usual care.

In addition to the primary aims, secondary outcomes will also be evaluated. The intervention is expected to enhance subjective and objective indices of fitness, increase quality of life, improve indices of diabetes management and decrease depression symptoms. Predictors of response to treatment will also be evaluated.

Results from this pilot study will be instrumental for guiding a subsequent, larger and longer term randomized study for evaluating reinforcement interventions for improving outcomes of youth and young adults with T1D.

ELIGIBILITY:
Inclusion Criteria:

* age 13-24 years old and live with a parent at least 4 days per week on average;
* diagnosis of type 1 diabetes >12 months via ADA guidelines;
* mean A1c>7.5% and <13% in the year before study entry, and most recent A1c >7.5% but <13%;
* check blood sugar at least 2 times per day on average;
* access to a computer or cell phone with Internet for uploading or synching activity monitoring data and text messaging or email capabilities to communicate with study staff
* currently walk at least 1,000 steps per day, but less than 6,000 steps per day on average as assessed on >11 days between baseline session 1 and baseline session 2
* English speaking, pass an informed consent quiz, and adequate knowledge of managing T1D

Exclusion Criteria:

* have a major psychiatric or neurocognitive disorder (e.g., severe learning impairment) or major visual impairment that would inhibit participation
* have a significant other medical condition that impacts diabetes management (e.g., eating disorder, rheumatoid arthritis, or other condition that requires steroid treatment) or a physical illness, injury or condition that may interfere with physical activity recommendations (e.g., joint, hip or back problems, uncontrolled hypertension, or BMI > 40 kg/m2)
* plan to switch insulin delivery mode (injection to pump or vice versa) in the next 6 months, or have recently switched
* participating in another clinical trial
* fail or is unable to upload or synch the activity meter at least 4 times during the baseline period

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
proportion of days participants walked the recommended number of steps | 12 weeks
  The proportion of days participants walked the recommended number of steps which the recommended number of steps was achieved on at least 5 of the 7 days.
proportion of days in the month participants walked 10,000 or more steps | 24 weeks
  Long-term outcome will be proportion of days in the month before the 24-week follow up on which participants walked 10,000 or more steps.
number of consecutive weeks step goal met | 12 weeks
  The number of weeks in a row in which the recommended number of steps was achieved on at least 5 of the 7 days.

SECONDARY OUTCOMES:
proportion of days participants walked the recommended number of steps | Baseline
  The proportion of days participants walked the recommended number of steps which the recommended number of steps was achieved on at least 5 of the 7 days.
proportion of days participants walked the recommended number of steps | 6 weeks
  The proportion of days participants walked the recommended number of steps which the recommended number of steps was achieved on at least 5 of the 7 days.
proportion of days participants walked the recommended number of steps | 24 weeks
  The proportion of days participants walked the recommended number of steps which the recommended number of steps was achieved on at least 5 of the 7 days.
proportion of days in the month participants walked 10,000 or more steps | Baseline
  The proportion of days participants walked the recommended number of steps which the recommended number of steps was achieved on at least 5 of the 7 days.
proportion of days in the month participants walked 10,000 or more steps | 6 weeks
  The proportion of days participants walked the recommended number of steps which the recommended number of steps was achieved on at least 5 of the 7 days.
proportion of days in the month participants walked 10,000 or more steps | 12 weeks
  The proportion of days participants walked the recommended number of steps which the recommended number of steps was achieved on at least 5 of the 7 days.
Body Mass Index | Baseline
  Body mass index (BMI) will be used as an indicator of physical activity and fitness. BMI will be calculated from height (assessed in stocking feet and measured to the nearest 0.10 cm) and weight (with excessive clothing, keys, wallets etc removed) and measured to the nearest 0.10 kg. BMI is weight in kg/height in m2. BMI range of > 0 to 40kg/m2. Higher BMI is perceived as unhealthy.
Body Mass Index | 6 weeks
  Body mass index (BMI) will be used as an indicator of physical activity and fitness. BMI will be calculated from height (assessed in stocking feet and measured to the nearest 0.10 cm) and weight (with excessive clothing, keys, wallets etc removed) and measured to the nearest 0.10 kg. BMI is weight in kg/height in m2. BMI range of > 0 to 40kg/m2. Higher BMI is perceived as unhealthy.
Body Mass Index | 12 weeks
  Body mass index (BMI) will be used as an indicator of physical activity and fitness. BMI will be calculated from height (assessed in stocking feet and measured to the nearest 0.10 cm) and weight (with excessive clothing, keys, wallets etc removed) and measured to the nearest 0.10 kg. BMI is weight in kg/height in m2. BMI range of > 0 to 40kg/m2. Higher BMI is perceived as unhealthy.
Body Mass Index | 24 weeks
  Body mass index (BMI) will be used as an indicator of physical activity and fitness. BMI will be calculated from height (assessed in stocking feet and measured to the nearest 0.10 cm) and weight (with excessive clothing, keys, wallets etc removed) and measured to the nearest 0.10 kg. BMI is weight in kg/height in m2. BMI range of > 0 to 40kg/m2. Higher BMI is perceived as unhealthy.
Waist Circumference | Baseline
  Waist circumference (WC) will be used as an indicator of physical activity and fitness. WC is measured at the height of the iliac crest with a Gulick tape measure to the nearest cm. Range is not applicable, but circumference will be > 0. A higher waist circumference is perceived as a negative outcome.
Waist Circumference | 6 weeks
  Waist circumference (WC) will be used as an indicator of physical activity and fitness. WC is measured at the height of the iliac crest with a Gulick tape measure to the nearest cm. Range is not applicable, but circumference will be > 0. A higher waist circumference is perceived as a negative outcome.
Waist Circumference | 12 weeks
  Waist circumference (WC) will be used as an indicator of physical activity and fitness. WC is measured at the height of the iliac crest with a Gulick tape measure to the nearest cm. Range is not applicable, but circumference will be > 0. A higher waist circumference is perceived as a negative outcome.
Waist Circumference | 24 weeks
  Waist circumference (WC) will be used as an indicator of physical activity and fitness. WC is measured at the height of the iliac crest with a Gulick tape measure to the nearest cm. Range is not applicable, but circumference will be > 0. A higher waist circumference is perceived as a negative outcome.
Systolic Blood Pressure | Baseline
  Systolic blood pressure (SBP) will be used as an indicator of physical activity and fitness. SBP (mmHg) will be taken in seated position using a semi-automated noninvasive BP unit (e.g., Suntech, Raleigh, NC). After 5 min of seated rest, BP will be taken twice, 2 minutes apart in the non-dominant arm until two consecutive readings are within 5 mmHg and averaged. Range is not applicable, but reading will be > 0. Higher SBP values are perceived as negative.
Systolic Blood Pressure | 6 weeks
  Systolic blood pressure (SBP) will be used as an indicator of physical activity and fitness. SBP (mmHg) will be taken in seated position using a semi-automated noninvasive BP unit (e.g., Suntech, Raleigh, NC). After 5 min of seated rest, BP will be taken twice, 2 minutes apart in the non-dominant arm until two consecutive readings are within 5 mmHg and averaged. Range is not applicable, but reading will be > 0. Higher SBP values are perceived as negative.
Systolic Blood Pressure | 12 weeks
  Systolic blood pressure (SBP) will be used as an indicator of physical activity and fitness. SBP (mmHg) will be taken in seated position using a semi-automated noninvasive BP unit (e.g., Suntech, Raleigh, NC). After 5 min of seated rest, BP will be taken twice, 2 minutes apart in the non-dominant arm until two consecutive readings are within 5 mmHg and averaged. Range is not applicable, but reading will be > 0. Higher SBP values are perceived as negative.
Systolic Blood Pressure | 24 weeks
  Systolic blood pressure (SBP) will be used as an indicator of physical activity and fitness. SBP (mmHg) will be taken in seated position using a semi-automated noninvasive BP unit (e.g., Suntech, Raleigh, NC). After 5 min of seated rest, BP will be taken twice, 2 minutes apart in the non-dominant arm until two consecutive readings are within 5 mmHg and averaged. Range is not applicable, but reading will be > 0. Higher SBP values are perceived as negative.
Diastolic Blood Pressure | Baseline
  Diastolic blood pressure (DBP) will be used as an indicator of physical activity and fitness. DBP (mmHg) will be taken in seated position using a semi-automated noninvasive BP unit (e.g., Suntech, Raleigh, NC). After 5 min of seated rest, BP will be taken twice, 2 minutes apart in the non-dominant arm until two consecutive readings are within 5 mmHg and averaged. Longer distance in meters walked is perceived as good. Range is not applicable, but reading will be > 0. High DBP values are perceived as negative.
Diastolic Blood Pressure | 6 weeks
  Diastolic blood pressure (DBP) will be used as an indicator of physical activity and fitness. DBP (mmHg) will be taken in seated position using a semi-automated noninvasive BP unit (e.g., Suntech, Raleigh, NC). After 5 min of seated rest, BP will be taken twice, 2 minutes apart in the non-dominant arm until two consecutive readings are within 5 mmHg and averaged. Longer distance in meters walked is perceived as good. Range is not applicable, but reading will be > 0. High DBP values are perceived as negative.
Diastolic Blood Pressure | 12 weeks
  Diastolic blood pressure (DBP) will be used as an indicator of physical activity and fitness. DBP (mmHg) will be taken in seated position using a semi-automated noninvasive BP unit (e.g., Suntech, Raleigh, NC). After 5 min of seated rest, BP will be taken twice, 2 minutes apart in the non-dominant arm until two consecutive readings are within 5 mmHg and averaged. Longer distance in meters walked is perceived as good. Range is not applicable, but reading will be > 0. High DBP values are perceived as negative.
Diastolic Blood Pressure | 24 weeks
  Diastolic blood pressure (DBP) will be used as an indicator of physical activity and fitness. DBP (mmHg) will be taken in seated position using a semi-automated noninvasive BP unit (e.g., Suntech, Raleigh, NC). After 5 min of seated rest, BP will be taken twice, 2 minutes apart in the non-dominant arm until two consecutive readings are within 5 mmHg and averaged. Longer distance in meters walked is perceived as good. Range is not applicable, but reading will be > 0. High DBP values are perceived as negative.
Six Minute Walk Test | 12 weeks
  The six minute walk test (SMWT) will be used as an indicator of physical activity and fitness. SMWT records distance (in meters) that patients cover when walking indoors at their own pace for 6 min, timed by a standard stopwatch. Range is not applicable, but time will be > 0. Higher SMWT values are perceived as positive/good.
Sit to Stand Test | 12 weeks
  The sit to stand test will be used as an indicator of physical activity and fitness. In the sit to stand test, the patient starts in a standing position and moves to the floor with buttocks to the ground and returns to standing as quickly as possible. Times (in seconds) from standing to standing, and from floor sitting to standing, are recorded, with best of 2 trials used. Range is not applicable, but time will be > 0. Higher scores are perceived as poor outcomes.
Harvard Step Test | Baseline
  The modified Harvard Step Test will be used as an indicator of physical activity and fitness. After 5 min of rest, participants will be asked to step onto and down from a step 30 cm (11.8 inches) in height for 3 minutes at a rate of 30 steps per minute. Heart rate will be measured for 30 seconds at 1, 2 and 3 minutes after completion of stepping. A Physical Fitness Score [(duration of exercise in seconds x 100) / (sum of the three heart rates)] will be computed. Heart rate will be measured at 1, 2 and 3 minutes after completion of stepping. Harvard Step Test score = (duration of exercise in seconds x 100) / (sum of the three heart rates). Range is not applicable, but scores will be >0. Higher scores are perceived as good.
Harvard Step Test | 6 weeks
  The modified Harvard Step Test will be used as an indicator of physical activity and fitness. After 5 min of rest, participants will be asked to step onto and down from a step 30 cm (11.8 inches) in height for 3 minutes at a rate of 30 steps per minute. Heart rate will be measured for 30 seconds at 1, 2 and 3 minutes after completion of stepping. A Physical Fitness Score [(duration of exercise in seconds x 100) / (sum of the three heart rates)] will be computed. Heart rate will be measured at 1, 2 and 3 minutes after completion of stepping. Harvard Step Test score = (duration of exercise in seconds x 100) / (sum of the three heart rates). Range is not applicable, but scores will be >0. Higher scores are perceived as good.
Harvard Step Test | 12 weeks
  The modified Harvard Step Test will be used as an indicator of physical activity and fitness. After 5 min of rest, participants will be asked to step onto and down from a step 30 cm (11.8 inches) in height for 3 minutes at a rate of 30 steps per minute. Heart rate will be measured for 30 seconds at 1, 2 and 3 minutes after completion of stepping. A Physical Fitness Score [(duration of exercise in seconds x 100) / (sum of the three heart rates)] will be computed. Heart rate will be measured at 1, 2 and 3 minutes after completion of stepping. Harvard Step Test score = (duration of exercise in seconds x 100) / (sum of the three heart rates). Range is not applicable, but scores will be >0. Higher scores are perceived as good.
Harvard Step Test | 24 weeks
  The modified Harvard Step Test will be used as an indicator of physical activity and fitness. After 5 min of rest, participants will be asked to step onto and down from a step 30 cm (11.8 inches) in height for 3 minutes at a rate of 30 steps per minute. Heart rate will be measured for 30 seconds at 1, 2 and 3 minutes after completion of stepping. A Physical Fitness Score [(duration of exercise in seconds x 100) / (sum of the three heart rates)] will be computed. Heart rate will be measured at 1, 2 and 3 minutes after completion of stepping. Harvard Step Test score = (duration of exercise in seconds x 100) / (sum of the three heart rates). Range is not applicable, but scores will be >0. Higher scores are perceived as good.
Physical Activity Questionnaire | Baseline
  The International Physical Activity Questionnaire, Short Form (IPAQ) will be used as an indicator of physical activity and fitness. IPAQ assesses total physical activity in the previous 7 days. Questions measure the frequency (days per week) and duration (minutes per session) of physical activity, as well as its intensity level (vigorous, moderate, walking, or sitting). Participants are categorized into one of three physical activity levels (low, moderate, high) using algorithms provided in the IPAQ short form scoring protocol (www.ipaq.ki.se). Range is not applicable because it is a categorical variable. The high activity category is perceived as good.
Physical Activity Questionnaire | 6 weeks
  The International Physical Activity Questionnaire, Short Form (IPAQ) will be used as an indicator of physical activity and fitness. IPAQ assesses total physical activity in the previous 7 days. Questions measure the frequency (days per week) and duration (minutes per session) of physical activity, as well as its intensity level (vigorous, moderate, walking, or sitting). Participants are categorized into one of three physical activity levels (low, moderate, high) using algorithms provided in the IPAQ short form scoring protocol (www.ipaq.ki.se). Range is not applicable because it is a categorical variable. The high activity category is perceived as good.
Physical Activity Questionnaire | 12 weeks
  The International Physical Activity Questionnaire, Short Form (IPAQ) will be used as an indicator of physical activity and fitness. IPAQ assesses total physical activity in the previous 7 days. Questions measure the frequency (days per week) and duration (minutes per session) of physical activity, as well as its intensity level (vigorous, moderate, walking, or sitting). Participants are categorized into one of three physical activity levels (low, moderate, high) using algorithms provided in the IPAQ short form scoring protocol (www.ipaq.ki.se). Range is not applicable because it is a categorical variable. The high activity category is perceived as good.
Physical Activity Questionnaire | 24 weeks
  The International Physical Activity Questionnaire, Short Form (IPAQ) will be used as an indicator of physical activity and fitness. IPAQ assesses total physical activity in the previous 7 days. Questions measure the frequency (days per week) and duration (minutes per session) of physical activity, as well as its intensity level (vigorous, moderate, walking, or sitting). Participants are categorized into one of three physical activity levels (low, moderate, high) using algorithms provided in the IPAQ short form scoring protocol (www.ipaq.ki.se). Range is not applicable because it is a categorical variable. The high activity category is perceived as good.
Habitual Total Weekend Activity Score | Baseline
  Habitual Activity Estimation Scale (HAES) will be used as an indicator of physical activity and fitness. The HAES asks participants to break their day down into four time periods; wakeup to breakfast, end of breakfast to lunch, end of lunch to supper, and end of supper to bedtime and to breakdown the activity done in each time period into; inactive, somewhat inactive, somewhat active, and very active. The HAES is filled out for both a typical weekday and weekend day. Total number of hours per day spent in each of four activity categories (inactive, somewhat inactive, somewhat active, and very active) will be calculated. Total activity (hours per day somewhat active + hours per day very active) also will be calculated. Two total activity scores are calculated - 1 for the weekday and 1 for the weekend day. Total activity score = hours per day somewhat active + hours per day very active.Total activity range of 0 to 24. High total activity is perceived as good.
Habitual Total Weekend Activity Score | 6 weeks
  Habitual Activity Estimation Scale (HAES) will be used as an indicator of physical activity and fitness. The HAES asks participants to break their day down into four time periods; wakeup to breakfast, end of breakfast to lunch, end of lunch to supper, and end of supper to bedtime and to breakdown the activity done in each time period into; inactive, somewhat inactive, somewhat active, and very active. The HAES is filled out for both a typical weekday and weekend day. Total number of hours per day spent in each of four activity categories (inactive, somewhat inactive, somewhat active, and very active) will be calculated. Total activity (hours per day somewhat active + hours per day very active) also will be calculated. Two total activity scores are calculated - 1 for the weekday and 1 for the weekend day. Total activity score = hours per day somewhat active + hours per day very active.Total activity range of 0 to 24. High total activity is perceived as good.
Habitual Total Weekend Activity Score | 12 weeks
  Habitual Activity Estimation Scale (HAES) will be used as an indicator of physical activity and fitness. The HAES asks participants to break their day down into four time periods; wakeup to breakfast, end of breakfast to lunch, end of lunch to supper, and end of supper to bedtime and to breakdown the activity done in each time period into; inactive, somewhat inactive, somewhat active, and very active. The HAES is filled out for both a typical weekday and weekend day. Total number of hours per day spent in each of four activity categories (inactive, somewhat inactive, somewhat active, and very active) will be calculated. Total activity (hours per day somewhat active + hours per day very active) also will be calculated. Two total activity scores are calculated - 1 for the weekday and 1 for the weekend day. Total activity score = hours per day somewhat active + hours per day very active.Total activity range of 0 to 24. High total activity is perceived as good.
Habitual Total Weekend Activity Score | 24 weeks
  Habitual Activity Estimation Scale (HAES) will be used as an indicator of physical activity and fitness. The HAES asks participants to break their day down into four time periods; wakeup to breakfast, end of breakfast to lunch, end of lunch to supper, and end of supper to bedtime and to breakdown the activity done in each time period into; inactive, somewhat inactive, somewhat active, and very active. The HAES is filled out for both a typical weekday and weekend day. Total number of hours per day spent in each of four activity categories (inactive, somewhat inactive, somewhat active, and very active) will be calculated. Total activity (hours per day somewhat active + hours per day very active) also will be calculated. Two total activity scores are calculated - 1 for the weekday and 1 for the weekend day. Total activity score = hours per day somewhat active + hours per day very active.Total activity range of 0 to 24. High total activity is perceived as good.
Habitual Total Weekday Activity Score | Baseline
  Habitual Activity Estimation Scale (HAES) will be used as an indicator of physical activity and fitness. The HAES asks participants to break their day down into four time periods; wakeup to breakfast, end of breakfast to lunch, end of lunch to supper, and end of supper to bedtime and to breakdown the activity done in each time period into; inactive, somewhat inactive, somewhat active, and very active. The HAES is filled out for both a typical weekday and weekend day. Total number of hours per day spent in each of four activity categories (inactive, somewhat inactive, somewhat active, and very active) will be calculated. Total activity (hours per day somewhat active + hours per day very active) also will be calculated. Two total activity scores are calculated - 1 for the weekday and 1 for the weekend day. Total activity score = hours per day somewhat active + hours per day very active.Total activity range of 0 to 24. High total activity is perceived as good.
Habitual Total Weekday Activity Score | 6 weeks
  Habitual Activity Estimation Scale (HAES) will be used as an indicator of physical activity and fitness. The HAES asks participants to break their day down into four time periods; wakeup to breakfast, end of breakfast to lunch, end of lunch to supper, and end of supper to bedtime and to breakdown the activity done in each time period into; inactive, somewhat inactive, somewhat active, and very active. The HAES is filled out for both a typical weekday and weekend day. Total number of hours per day spent in each of four activity categories (inactive, somewhat inactive, somewhat active, and very active) will be calculated. Total activity (hours per day somewhat active + hours per day very active) also will be calculated. Two total activity scores are calculated - 1 for the weekday and 1 for the weekend day. Total activity score = hours per day somewhat active + hours per day very active.Total activity range of 0 to 24. High total activity is perceived as good.
Habitual Total Weekday Activity Score | 12 weeks
  Habitual Activity Estimation Scale (HAES) will be used as an indicator of physical activity and fitness. The HAES asks participants to break their day down into four time periods; wakeup to breakfast, end of breakfast to lunch, end of lunch to supper, and end of supper to bedtime and to breakdown the activity done in each time period into; inactive, somewhat inactive, somewhat active, and very active. The HAES is filled out for both a typical weekday and weekend day. Total number of hours per day spent in each of four activity categories (inactive, somewhat inactive, somewhat active, and very active) will be calculated. Total activity (hours per day somewhat active + hours per day very active) also will be calculated. Two total activity scores are calculated - 1 for the weekday and 1 for the weekend day. Total activity score = hours per day somewhat active + hours per day very active.Total activity range of 0 to 24. High total activity is perceived as good.
Habitual Total Weekday Activity Score | 24 weeks
  Habitual Activity Estimation Scale (HAES) will be used as an indicator of physical activity and fitness. The HAES asks participants to break their day down into four time periods; wakeup to breakfast, end of breakfast to lunch, end of lunch to supper, and end of supper to bedtime and to breakdown the activity done in each time period into; inactive, somewhat inactive, somewhat active, and very active. The HAES is filled out for both a typical weekday and weekend day. Total number of hours per day spent in each of four activity categories (inactive, somewhat inactive, somewhat active, and very active) will be calculated. Total activity (hours per day somewhat active + hours per day very active) also will be calculated. Two total activity scores are calculated - 1 for the weekday and 1 for the weekend day. Total activity score = hours per day somewhat active + hours per day very active.Total activity range of 0 to 24. High total activity is perceived as good.

CONTACTS AND LOCATIONS:
Overall Officials: William Tamborlane, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No